CLINICAL TRIAL: NCT06665464
Title: Bioavailability of Omega-3 Fatty Acids From Fish Oil Supplements
Acronym: Ocean's O3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wageningen University and Research (Other)
Responsible Party: Principal Investigator, Lonneke Janssen Duijghuijsen, Researcher Clinical Trials, Wageningen University and Research
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: NL87485.041.24
Record Dates: First submitted 2024-10-29; First posted 2024-10-30 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Nutrition; Absorption, Metabolism and Excretion in Healthy Volunteers; Fish Oils; Omega 3 Fatty Acids
Keywords: Omega 3 fatty acids; bioavailability; oral supplement; fish oil supplement

STUDY DESIGN:
Intervention Model Description: This intervention study has a randomized, cross-over, open label design
Masking Description: The researchers performing the sample and data analyses will be blinded until all analyses are finalized.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fish oil supplement 1 (Active Comparator)
  Interventions: Dietary Supplement: Fish oil supplement 1
- Fish oil supplement 2 (Experimental)
  Interventions: Dietary Supplement: Fish oil supplement 2

INTERVENTIONS:
Dietary Supplement: Fish oil supplement 1 — Soft gel capsule
  Arms: Fish oil supplement 1
Dietary Supplement: Fish oil supplement 2 — Soft gel chewable
  Arms: Fish oil supplement 2

SUMMARY:
This study is investigating whether a new type of fish oil supplement, in the form of soft chews, leads to better absorption of omega-3s in the body compared to traditional fish oil capsules. Omega-3s, found in fish oil, are known to support heart health and reduce inflammation, but they may absorb better in certain forms. In this study, participants will take both types of supplements (soft chews and capsules) at different times to compare how well the omega-3s are absorbed. Researchers will measure the levels of omega-3s in the blood over several hours to determine if the soft chews offer a better option for people seeking the health benefits of omega-3s.

ELIGIBILITY:
Inclusion Criteria:

* Apparently healthy adults (18 - 50 yrs);
* Body mass index (BMI) ≥18.5 and ≤30 kg/m2;
* Having veins suitable for blood sampling via a catheter (judged by study nurse/ medical doctor);
* Willing to refrain from fish, fish oil, and products with added omega-3 starting from 2 weeks prior to the first postprandial test day and during the study period;
* Willing to keep a stable dietary pattern throughout the study.

Exclusion Criteria:

* Having a disease that may interfere with the outcomes of this study, such as a known metabolic, gastrointestinal, inflammatory or chronic disease (such as anaemia, diabetes, hepatitis, hypercholesterolemia, cardiovascular disease), as judged by the medical investigator.
* Having a history of medical or surgical events that may significantly affect the study outcome, including: inflammatory bowel disease, pancreatitis, ulcers, gastrointestinal or rectal bleeding; major gastrointestinal tract surgery such as gastrectomy, gastroenterostomy, or bowel resection; known or suspected gastrointestinal disorders, colon or GI tract cancer;
* Use of medication that may interfere with the study outcomes, including gastric acid inhibitors, laxatives, and lipid lowering drugs, as judged by the medical supervisor;
* Anaemia (Haemoglobin (Hb) values <7.5 mmol/L for women and <8.5 mmol/L for men), as assessed by finger prick blood during screening visit; NL87485.041.24 Ocean's O3
* Allergic for fish;
* Having swallowing problems with capsules;
* Recent blood donation (<1 month prior to test day 1 of the study) or not willing to stop donation during and 1 month after the study;
* Average alcohol intake >21 (women) or >28 (men) glasses of alcoholic beverages per week;
* Reported to follow or having planned a slimming or medically prescribed diet;
* Use of recreational drugs;
* Current smokers, or stopped smoking in the last 3 months before study start;
* Insufficient proficiency in Dutch to understand information brochure and questionnaires
* Participation in any clinical trial including blood sampling and/or administration of substances up to 30 days before test day 1 of this study and during the study period;
* Being an employee of the department Food, Health & Consumer Research Wageningen Food & Biobased Research.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2024-11-20 (Actual); Primary Completion 2024-12-19 (Actual); Study Completion 2024-12-19 (Actual)

PRIMARY OUTCOMES:
The area under the curve of combined EPA and DHA plasma levels in venous blood samples | Between baseline and 24 hours
  Venous blood samples collected at baseline (t=-15min and t=0) and at t=30, 60, 90, 120, 150, 180, 240, 360, 540, and 720min, and 24hours

SECONDARY OUTCOMES:
The time to peak for combined EPA and DHA plasma levels | Between baseline and 24 hours
  Venous blood samples collected at baseline (t=-15min and t=0) and at t=30, 60, 90, 120, 150, 180, 240, 360, 540, and 720min, and 24hours
The maximum peak height for combined EPA and DHA plasma levels | Between baseline and 24 hours
  Venous blood samples collected at baseline (t=-15min and t=0) and at t=30, 60, 90, 120, 150, 180, 240, 360, 540, and 720min, and 24hours
The area under the curve of DHA plasma levels in venous blood samples | Between baseline and 24 hours
  Venous blood samples collected at baseline (t=-15min and t=0) and at t=30, 60, 90, 120, 150, 180, 240, 360, 540, and 720min, and 24hours
The area under the curve of EPA plasma levels in venous blood samples | Between baseline and 24 hours
  Venous blood samples collected at baseline (t=-15min and t=0) and at t=30, 60, 90, 120, 150, 180, 240, 360, 540, and 720min, and 24hours
The time to peak for DHA plasma levels | Between baseline and 24 hours
  Venous blood samples collected at baseline (t=-15min and t=0) and at t=30, 60, 90, 120, 150, 180, 240, 360, 540, and 720min, and 24hours
The time to peak for EPA plasma levels | Between baseline and 24 hours
  Venous blood samples collected at baseline (t=-15min and t=0) and at t=30, 60, 90, 120, 150, 180, 240, 360, 540, and 720min, and 24hours
The maximum peak height for EPA plasma levels | Between baseline and 24 hours
  Venous blood samples collected at baseline (t=-15min and t=0) and at t=30, 60, 90, 120, 150, 180, 240, 360, 540, and 720min, and 24hours
The maximum peak height for DHA plasma levels | Between baseline and 24 hours
  Venous blood samples collected at baseline (t=-15min and t=0) and at t=30, 60, 90, 120, 150, 180, 240, 360, 540, and 720min, and 24hours

CONTACTS AND LOCATIONS:
Locations (1):
- Wageningen University & Research, Wageningen, Netherlands

IPD SHARING:
Plan to Share IPD: No
No consent from study participants